CLINICAL TRIAL: NCT03240016
Title: ABLE: Phase II, Single Arm, Two-stage Study of Abraxane With Anti-PD1/PDL1 in Patients With Advanced Urothelial Cancer
Brief Title: Abraxane With Anti-PD1/PDL1 in Patients With Advanced Urothelial Cancer
Acronym: ABLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.077; HUM00135166 (Other: University of Michigan)
Record Dates: First submitted 2017-07-27; First posted 2017-08-04 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab and Abraxane (Experimental): Pembrolizumab 200mg IV D1 Abraxane 100mg/m^2 IV D1 and D8 21 Day Cycles
  Interventions: Drug: Pembrolizumab; Drug: Abraxane

INTERVENTIONS:
Drug: Pembrolizumab — 200mg IV D1
Drug: Abraxane — 100mg/m^2 D1 and D8

SUMMARY:
This is a phase 2, single arm, two-stage study of abraxane with an anti-PD1/PDL1 (pembrolizumab) in cisplatin-ineligible patients with advanced urothelial cancer.

Each cycle last 21-days. All subjects will receive pembrolizumab via IV on day 1, and abraxane via IV on Day 1 and Day 8 of each cycle. Subjects may continue to receive the study regimen until they experience disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent unresectable locally advanced or metastatic urothelial carcinoma (aka transitional cell carcinoma).
* Patients may be either cisplatin-ineligible or platinum-refractory.
* Histological or cytologically proven urothelial carcinoma.
* Have measurable disease based on RECIST 1.1
* Has urothelial cancer that is not suitable for local therapy administered with curative intent if not already administered.
* Must have recovered (i.e., AE <= Grade 1 or stable) from AEs due to a previously administered agent.
* ECOG Performance Status of 0, 1 or 2. (Eastern Cooperative Oncology Group Performance Status: an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.)
* Prior neoadjuvant or adjuvant systemic therapy or local intravesical chemotherapy or immunotherapy is permitted.
* Adequate organ and marrow function
* Women of child-bearing potential must either commit to true abstinence or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting IP therapy, and while on study medication or for a longer period if required by local regulations following the last dose of IP; and have a negative serum pregnancy test result at screening
* Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following drug discontinuation, even if he has undergone a successful vasectomy.
* Patients must have < Grade 2 pre-existing peripheral neuropathy
* Be ≥18 years of age as of date of signing informed consent
* Voluntarily agree to participate by providing written informed consent/assent for the trial

Exclusion Criteria:

* Prior exposure to immune-mediated therapy
* History of allogenic organ transplantation that requires ongoing use of immunosuppressive agents is NOT permitted
* Active or prior documented autoimmune or inflammatory disorders are NOT permitted
* Current or prior use of immunosuppressive medication(s) within 14 days before study treatment is NOT permitted.
* Brain metastases or spinal cord compression are NOT permitted unless they have been treated with the patient's condition being stable clinically and radiologically for 28 calendar days and off steroids for at least 14 days prior to the start of study treatment.
* Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) is NOT permitted.
* Receipt of live attenuated vaccine within 30 days prior to the first study treatment is NOT permitted.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 28 calendar days of the first dose of treatment.
* CTCAE Grade > 1 peripheral neuropathy is NOT permitted
* If subjects received major surgery they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting trial therapy
* Has a known additional malignancy that is progressing or requires active treatment
* Has a history of severe hypersensitivity reaction to nab-paclitaxel or anti-PD1/PDL1
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnancies:

  1. Females: nab-paclitaxel can cause harm to an unborn child if given to a pregnant woman. Females may not take part in this study if pregnant or breast-feeding for 6 months after last dose of study drug.
  2. Males: Male subjects should avoid fathering a child while receiving study medication and for 6 months after the last dose of study medication. Males must agree to complete abstinence from heterosexual contact or use a condom during sexual contact with a female of child bearing potential while receiving study medication and within 6 months after last dose of study medication.
  3. Subjects (both males and female) should practice effective contraception during study and for 6 months after the last dose of study medication (Section 3.1.8 i, ii).
* Patients with biliary obstruction or biliary stent are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajjai Alva, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Tsung I, Green E, Palmbos P, Sloan Z, Reichert ZR, Vaishampayan U, Smith DC, Caram MEV, Yentz S, Daignault-Newton S, Hurley L, Nguyen CB, Kraft S, Alva A. A Phase 2 Trial of Nab-paclitaxel in Combination With Anti-PD1 Therapy in Advanced Urothelial Cancer. J Urol. 2023 Jan;209(1):121-130. doi: 10.1097/JU.0000000000002969. Epub 2022 Nov 1. PMID 36317715

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab and Abraxane
Started | 36
Completed | 17
Not Completed | 19
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 7
Not completed — Death | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and Abraxane
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients That Respond to Treatment
Description: The Overall Response Rate (ORR) will be the percentage of patients that achieve either complete response (CR) or partial response (PR).
  CR is defined as the disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
  PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
Time Frame: 24 months post treatment, an average of 7.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab and Abraxane
Number analyzed (Participants) | 36
Participants | 18

2. Secondary Outcome: Duration of Response
Description: The duration of response (DOR) is measured from the time that response (PR or CR) criteria are met until the first date that recurrent or progressive disease is objectively documented.
  CR is defined as the disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
  PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
Time Frame: 24 months post treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab and Abraxane
Number analyzed (Participants) | 18
months | 4.4 [4.0 to 8.6]

3. Secondary Outcome: Progression Free Survival Time
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death.
  Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: 24 months post treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab and Abraxane
Number analyzed (Participants) | 36
months | 6.8 [4.4 to NA] — not reached

4. Secondary Outcome: Median Number of Patients Alive at 12 and 24 Months
Description: Overall survival will be documented as the median number of patients alive at 12 and 24 months.
Time Frame: 12 and 24 months post treatment
Measure: Number (95% Confidence Interval); unit: binomial proportion of patients alive
Arm/Group | Pembrolizumab and Abraxane
Number analyzed (Participants) | 36
binomial proportion of patients alive
  12 Months | 0.83 [0.71 to 0.96]
  24 Months | 0.77 [0.64 to 0.91]

5. Secondary Outcome: Median Duration of Therapy
Time Frame: from the start of therapy, up to 24 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Pembrolizumab and Abraxane
Number analyzed (Participants) | 36
days | 157 [85 to 292]

6. Secondary Outcome: Percentage of Patients That Completely Respond to Treatment
Description: The percentage of patients that achieve complete response to treatment. Complete response is defined as the disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
Time Frame: 24 months post treatment, an average of 7.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab and Abraxane
Number analyzed (Participants) | 36
Participants | 3

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment. Up to 2 years.
Arm/Group | Pembrolizumab and Abraxane
All-Cause Mortality (participants affected / at risk) | 13/36
Serious Adverse Events (participants affected / at risk) | 17/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Abraxane (N=36)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — pyelonephritis
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — disease progression
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Transient ischemic attack/brain ischemia
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — hiccoughs
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — pneumonia
Sepsis (Infections and infestations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Abraxane (N=36)
Abdominal Pain (Gastrointestinal disorders) | 5 (6)
Acute kidney injury (Renal and urinary disorders) | 5 (5)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alopecia (General disorders) | 6 (6)
Anemia (Investigations) | 8 (13)
Anorexia (Metabolism and nutrition disorders) | 3 (6)
Arthralgia (General disorders) | 3 (4)
Arthritis (General disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Blurred vision (General disorders) | 4 (6)
Confusion (Psychiatric disorders) | 4 (6)
Constipation (Gastrointestinal disorders) | 5 (7)
Cough (General disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Dental caries (General disorders) | 2 (4)
Depression (Psychiatric disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Dizziness (General disorders) | 3 (3)
Dysarthria (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysgeusia (General disorders) | 5 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 3 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (7)
Fatigue (General disorders) | 14 (29)
Fever (General disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (4)
Headache (Nervous system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 3 (8)
Hypertension (Vascular disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 4 (9)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (8)
Neutrophil count decreased (Investigations) | 2 (4)
Pain (General disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Paresthesia (Nervous system disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6)
Sepsis (Infections and infestations) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 4 (5)
Weight loss (Investigations) | 4 (6)
White blood cell decreased (Investigations) | 2 (4)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2) — dysuria

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT03240016/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT03240016/ICF_001.pdf